CLINICAL TRIAL: NCT06139185
Title: "ASSOCIATION BETWEEN NASAL SEPTUM DEVIATION AND ALLERGIC RHINITIS IN PEDIATRIC AGE: The ARHINASD (Allergic Rhinitis in Pediatric Subjects With Nasal Septum Deviation) Project"
Brief Title: The ARHINASD (Allergic Rhinitis in Pediatric Subjects With Nasal Septum Deviation) Project
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Medical Doctor, PhD, Professor, Federico II University
Other Study IDs: 31/23
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with nasal septum deviation
  Interventions: Other: Data collection
- Patients without nasal septum deviation
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
Allergic rhinitis is one of the most common inflammatory conditions of the upper airway mucosa, especially in the pediatric population with a prevalence of approximately 25%. It is among the most common chronic inflammatory diseases globally and is caused by IgE-mediated reactions to inhaled allergens, often co-occurring with asthma and causing severe burdens and disabilities worldwide. Allergic rhinitis can in fact seriously compromise the quality of life, significantly influencing school performance, social life and the quality of sleep. It is known that the most common symptoms characterizing allergic rhinitis (itching of the nose, sneezing, rhinorrhea and nasal/sinus obstruction) are partly overlapping with those due to a condition of deviation of the nasal septum and a recent study has shown how 87 % of patients with persistent allergic rhinitis are affected by at least 1 of the 7 types of nasal septum deformity. Deviation of the nasal septum is a very frequent anatomical disorder and is present in up to 48% of children and adolescents in the general population. The deviation narrows the affected nostril canal, reducing the flow of air that passes through the nostrils, predisposing to chronic mucosal inflammation with inflammatory infiltrate and in turn increasing the risk of developing chronic rhinitis and sinusitis. There are no data in the literature that correlate nasal septum deviation with an increased risk of developing allergic rhinitis. Given these premises, the ARHINASD (Allergic Rhinitis in pediatric topics with Nasal Septum Deviation) study was designed with the primary objective of evaluating the presence of allergic rhinitis in a sample of patients with and without deviation of the nasal septum.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity
* both sexes
* age between 6 and 14 years
* written informed consent.

Exclusion Criteria:

* Non-Caucasian ethnicity
* Age <6 and >14 years

Concomitant presence of:

* chronic diseases
* malignancies
* immunodeficiency
* chronic infections
* autoimmune diseases
* chronic inflammatory intestinal diseases
* celiac disease
* genetic diseases
* metabolic diseases
* cystic fibrosis
* chronic pulmonary diseases
* malformations of the cardiovascular system
* malformations of the respiratory system
* malformations of the gastrointestinal system
* neuropsychiatric disorders
* neurological diseases
* obesity
* eosinophilic diseases
* antibiotics use in the last 7 days
* cortisone use in the last 7 days
* antihistamines use in the last 7 days
* trauma at nose level in the 3 years before the enrollment,
* history of previous nose surgery, or previous major surgery procedures of gastrointestinal, cardiovascular, urinary or respiratory tract

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Caucasian children of both sexes aged between 6 and 14 with and without suspected deviation of the nasal septum observed at Pediatrics Section of Department of Translational Medical Sciences (University of Naples Federico II), University of Calabria (Department of Pharmacy, Health and Nutrition Sciences) and Otorhinolaryngology Unit, Penne Hospital, ASL of Pescara
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Presence of allergic rhinitis | 12 months
  Complete clinical and anamnestic evaluation and allergy screening test (Skin-Prick Test).

SECONDARY OUTCOMES:
Total IgE of nasal wash supernatant | 12 months
  ELISA kit
Cytokines (IL-13, IL-9, IL-33, IL-5, INFγ, β-defensin, IL-17, TNFα) of nasal wash supernatant | 12 months
  ELISA kit
Quality of life questionnaire | 12 months
  Quality of life questionnaire (VAS)
Peak inspiratory nasal flow | 12 months
  PNIF test
Nasal cytology | 12 months
  Performed with the nasal scraping to obtain cells which are then stained with May-Grunwald and Giemsa staining and observed using an optical microscope

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Department of Traslational Medical Science - University of Naples Federico II, Naples
  - University of Naples Federico II, Naples

IPD SHARING:
Plan to Share IPD: No